CLINICAL TRIAL: NCT01383122
Title: The Efficacy of Pulsed Electromagnetic Field Therapy for Management of Post-operative Pain Following Cesarean Delivery: a Randomised, Double-blind, Placebo-controlled Study
Brief Title: The Efficacy of Pulsed Electromagnetic Field Therapy for Management of Post-operative Pain Following Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Planned interim analysis-no statistical significance for the primary outcome.
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose C.A. Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-01
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Pain
Keywords: Pulsed electromagnetic field device; Cesarean section
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active device (Active Comparator): Functional pulsed electromagnetic field device
  Interventions: Device: Pulsed electromagnetic field device (ActiPatch TM)
- Placebo - inactive device (Placebo Comparator): Inactive pulsed electromagnetic field device
  Interventions: Device: Inactive pulsed electromagnetic field device (ActiPatch TM)

INTERVENTIONS:
Device: Pulsed electromagnetic field device (ActiPatch TM) — Wire loop of pulsed electromagnetic field device is taped around the wound for 48 hours.
  Other Names: ActiPatch TM
  Arms: Active device
Device: Inactive pulsed electromagnetic field device (ActiPatch TM) — Wire loop of pulsed electromagnetic field device is taped around the wound for 48 hours.
  Other Names: ActiPatch TM
  Arms: Placebo - inactive device

SUMMARY:
Pain following Cesarean delivery remains the most common post-operative complaint, and the provision of effective and safe analgesia is very important. Pain can impede the mother's ability to mobilise, and to care for and breastfeed her newborn baby.

Pulsed electromagnetic field (PEMF) devices have been used in various clinical settings, especially after plastic surgeries, to reduce postoperative swelling and pain, as well as to accelerate wound repair. PEMF therapy is simple to use, cost-effective and has no known side effects.

Despite advances in post-operative analgesia, pain relief and maternal satisfaction remain inadequate in some patients. Improving the quality of post-Cesarean analgesia while limiting undesirable side effects will enhance maternal satisfaction and reduce the risk of post-operative complications.

The investigators hypothesize that the continuous use of a PEMF device for 48 hours after Cesarean delivery will result in decreased post-operative pain scores on movement at 48 hours.

DETAILED DESCRIPTION:
Currently, at our institution, analgesic regimens are multimodal, in that they combine analgesic drugs with differing mechanisms of action, with the aim of producing effective analgesia while minimising adverse effects. They include opioid drugs, administered both neuro-axially and systemically, as well as paracetamol and non-steroidal anti-inflammatory drugs (NSAIDs). Opioids, while effective, have significant adverse effects, including sedation, nausea, vomiting and constipation. Non-steroidal anti-inflammatory drugs (NSAIDs) can reduce opioid consumption, but also have side effects, and are contra-indicated in a significant number of patients. Therefore there remains considerable scope to improve post-Cesarean analgesia.

Pulsed electromagnetic field (PEMF) technology relieves edema, inflammation and pain by stabilizing leaking cell membranes. The short bursts of electrical current do not produce heat or interfere with nerve or muscle function. The pulsed energy drives out edematous fluid along with by-products of the damaged tissue, which reduces swelling and helps re-establish cell-cell communication. The device is easily applied over the wound dressing, and has no known side effects for either the mother or the infant.

As the rate of Cesarean delivery continues to increase, and there remain significant problems with current analgesic regimens, the use of pulsed electromagnetic field therapy has the potential to considerably improve acute and chronic post-Cesarean pain management, and lead to a widespread change in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* full term singleton pregnancy
* undergoing elective cesarean delivery

Exclusion Criteria:

* Patients who have refused, are unable to give or have withdrawn consent
* Patients unable to communicate fluently in English
* Patients with American Society of Anesthesiologists (ASA) classification of 3 or greater
* Patients with chronic pain, or neuropathic analgesic drugs
* Patients in use of antidepressant and psychotropic drugs
* Patients with a history of opioid or intravenous drug abuse
* Patients with known allergy or contra-indication to any other drugs used in this trial
* Patients who have refused spinal anesthesia, or those in whom it is contra-indicated
* Patients with a history of previous cesarean delivery and persistent pain

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pain score by visual analogue scale (VAS) on movement at 48 hours postoperatively | 48 hours

SECONDARY OUTCOMES:
Pain at rest and on movement by VAS, and maternal satisfaction at 24 & 48 hours postoperatively | 48 hours
Opioid consumption at 24 & 48 hours postoperatively | 48 hours
Assessment of side effects: nausea, vomiting, sedation & itchiness | 48 hours
Presence of pain 6 weeks postoperatively | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021